CLINICAL TRIAL: NCT04693975
Title: Impact of Social Distancing During the COVID-19 Pandemic on Non-infected People With Chronic Respiratory Diseases
Brief Title: Social Distancing During the COVID-19 Pandemic and People Living With Chronic Respiratory Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Nídia A Hernandes, Principal Investigator, Universidade Estadual de Londrina
Other Study IDs: PIDS-PC
Record Dates: First submitted 2020-11-30; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Idiopathic Pulmonary Fibrosis; Asthma Chronic
Keywords: physical inactivity; sedentarism; chronic lung diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Idiopathic Pulmonary Fibrosis; Sedentary Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Social distancing during the COVID-19 pandemic could lead to clinical and functional deterioration of people living with chronic respiratory diseases (CRD). As they are considered risk group for COVID-19, it is not recommended that they leave their house and have interaction with people outside. Thus, most of them have not been attend Pulmonary Rehabilitation sections since the beginning of pandemic, neither exercising outdoor, experiencing drastic restrictions in their activities of daily living.

It is well known that low level of physical activity in daily life (PADL) in this population is related to poor prognosis, including higher chance of hospitalization due to exacerbation and mortality. Therefore, the aim of this study is to evaluate the short- and mid-term impact of the COVID-19 pandemic on the clinical, physical and functional conditions and the PADL level of people living with CRD (chronic obstructive pulmonary disease, asthma and interstitial lung diseases).

Participants will be assessed during the social isolation period and they will be reassessed immediately after release from social isolation. Thus, the subjects will be followed-up during 12 months to record symptoms, functional status, quality of life, exacerbations and hospitalizations.

The researchers' hypothesis is that those patients will present very low level of PADL in association to sedentarism, poor functional status, more symptoms of dyspnoea, anxiety and depression, poor sleep quality and, consequently, will present more episodes of acute exacerbation of the disease and more hospital admission during the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic obstructive pulmonary disease, asthma or interstitial lung disease;
* Absence of any severe and/or unstable cardiac disease;
* Absence of any orthopedic or neuromuscular condition that limits physical activity in daily life.

Exclusion Criteria:

* Desire to leave the study at any time;
* Infection with SARS-CoV-2 during the study protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects living with a chronic lung disease who are not infected with SARS-CoV-2.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Physical activity in daily life | 24 months
  The totality of voluntary movement produced by skeletal muscles during everyday functioning will be assess by an activity monitor (ActiGraph) which will provide data of number of steps per day, and time spent in postures and activities of different intensities.
Patient's perception of physical activity in daily life | 24 months
  The questionnaire PROactive Physical Activity in COPD, that measures the patients' percpetion of physical activities performed in daily living, will be used to complement the evaluation of physical activity level. It is composed by 12 items that evaluate difficulty in performing activities in daily life. Each item scores from 0 to 4; the total score is provided by summing all items and higher scores indicate higher physical activity level.

SECONDARY OUTCOMES:
Dyspnoea sensation in daily living | 24 months
  The Medical Research Council (MRC) scale will be used to assess limitation in activities of daily living due to dyspnoea sensation. The scale varies from 1 to 5 points; higher scores indicate higher limitation due to dyspnoea.
Acute exacerbation | 24 months
  Acute exacerbations are episodes of acute worsening of the respiratory symptoms of patients with chronic lung disease, that result in additional therapy. Occurrence of those episodes during the research protocol will be self-reported in the visits.
Hospitalization | 24 months
  Hospital admission due to respiratory conditions. Occurrence of this event during the research protocol will be self-reported in the visits.
Functional status | 24 months
  Functional status is an individual's ability to perform normal daily activities required to meet basic needs, fulfill usual roles, and maintain health and well-being. The London Chest Activity of Daily Living (LCADL) scale, a validated tool to assess patients with chronic pulmonary disease, will be used to assess functional limitation. The scale is composed by 15 items divided in 4 domains; each item is scored from 0 to 5 points, indicating to what extent dyspnoea sensation limits functionality. The total score is calculated by summing all items; higher scores indicate worse functional status.
Health-related Quality of life | 24 months
  Quality of life is a term used to refer to an individual's total well-being. An specific questionnaire, the Brazilian version of the Modified Saint George´s Respiratory Questionnaire (mSGRQ), will be used to assess those patients with COPD and asthma. It is composed by 50 items that evaluate limitation of quality of life due to respiratory symptoms; they are divided in 3 domains: symptoms, activity and impact. Patients' responses are "agree" or "do not agree". The total score is calculated by summing the 3 domains; higher scores indicate worse quality of life.
Health-related Quality of life | 24 months
  Quality of life is a term used to refer to an individual's total well-being. An specific questionnaire, the Brazilian version of the Saint George´s Respiratory Questionnaire specifically developed for idiopathic pulmonary fibrosis patients (SGRQ-I), will be used to assess those patients with interstitial lung diseases. It is composed by 34 items that evaluate limitation of quality of life due to respiratory symptoms; they are divided in 3 domains: symptoms, activity and impact. The total score is calculated by summing the 3 domains varing from 0 to 100; higher scores indicate more impaired quality of life.
Sleep quality | 24 months
  Sleep quality is defined as one's satisfaction of the sleep experience, integrating aspects of sleep initiation, sleep maintenance, sleep quantity, and refreshment upon awakening. The Pittsburgh Sleep Quality Index (PSQI) will be used to asssess sleep quality. It is composed by 19 item grouped into 7 components: sleep duration, sleep disturbance, sleep latency, daytime dysfunction due to sleepiness, sleep efficiency, overall sleep quality, sleep medication use. Each of the sleep components yields a score ranging from 0 to 3; the total score is provided by summing all components, ranging from 0 to 21 points with the higher total score indicating worse sleep quality.
Anxiety and depression | 24 months
  Presence of symptoms of anxiety and depression that the patients are experiencing will be assess by the Hospital Anxiety and Depression Scale (HADS). It is a 14-item scale with 7 items each for anxiety and depression subscales. Scoring for each item ranges from 0 to 3. A subscale score > 8 indicates anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Nidia A Hernandes, PhD, Principal Investigator — State University of Londrina
Locations (1):
- Laboratory of Reasearch in Respiratory Physiotherapy, State University of Londrina, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No